CLINICAL TRIAL: NCT05675280
Title: The Association Between Iron Deficiency at Diagnosis, Female Sex and Tissue Transglutaminase Antibody Normalization in Pediatric Celiac Disease
Brief Title: Iron Deficiency and TTG Normalization
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, eyal zifman, Head of pediatric gastroenterology service, Meir Medical Center
Other Study IDs: MMC-20-0021
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Celiac Disease in Children
MeSH Terms: interventions — Diet, Gluten-Free

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iron deficiency at diagnosis
  Interventions: Other: Gluten free diet
- No iron deficiency at diagnosis
  Interventions: Other: Gluten free diet

INTERVENTIONS:
Other: Gluten free diet — All subjects initiated a gluten free diet as mandated by their diagnosis of Celiac disease, regardless of the study

SUMMARY:
The investigators conducted a retrospective, observational cohort study which enrolled CD subjects aged 2-18y, diagnosed between Jan 2016 and Dec 2020. Demographic and laboratory data were collected at diagnosis and 1y after adherence to GFD. ID was determined according to hemoglobin and ferritin levels. The investigators compared CD subjects with and without ID at CD diagnosis in relation to TTG normalization at 1y.

ELIGIBILITY:
Inclusion Criteria:

* Children (male and female) diagnosed with CD
* Age 2-18y

Exclusion Criteria:

* Total IgA deficiency
* Anemia due to other causes - anyone with anemia and normal or elevated ferritin levels (e.g. thalassemia, spherocytosis)
* Other chronic conditions increasing the risk of anemia or falsely elevated ferritin (e.g. inflammatory bowel disease, chronic kidney disease, infection)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients diagnosed with Celiac disease
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
TTG normalization | 1 year from gluten free diet initiation
  normalization of tissue transglutaminase antibody

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Zifman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medical center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No